CLINICAL TRIAL: NCT01216293
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Dexlansoprazole 60 mg Delayed Release Capsules and Esomeprazole 40 mg Delayed Release Capsules on Bone Homeostasis in Healthy Postmenopausal Female Subjects
Brief Title: Effect of Dexlansoprazole on Bone Homeostasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-390MR_104; U1111-1116-1638 (Registry Identifier: WHO)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Homeostasis; Bone and Bones
Keywords: Drug Therapy
MeSH Terms: interventions — Dexlansoprazole; Lansoprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, once daily for up to 26 weeks. Participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 calcium (42 Ca) 3 milligram (mg), intravenously and 44 calcium (44 Ca) 8 mg, orally, once on Day-1 and Week 26.
  Interventions: Drug: Placebo
- Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg, capsules, orally, once daily for up to 26 weeks. Participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 Ca 3 mg, intravenously and 44 Ca 8 mg, orally, once on Day-1 and Week 26.
  Interventions: Drug: Dexlansoprazole
- Esomeprazole 40mg (Active Comparator): Esomeprazole 40 mg, capsules, orally, once daily for up to 26 weeks. Participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 Ca 3 mg, intravenously and 44 Ca 8 mg, orally, once on Day-1 and Week 26.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole 60 mg capsules
  Other Names: Dexilant; Kapidex
  Arms: Dexlansoprazole 60 mg
Drug: Esomeprazole — Esomeprazole 40 mg capsules
  Other Names: Nexium
  Arms: Esomeprazole 40mg
Drug: Placebo — Placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of dexlansoprazole modified release (MR), once daily (QD), on bone homeostasis.

DETAILED DESCRIPTION:
Research on drugs that affect bone homeostasis have shown changes in levels of bone formation and resorption biomarkers. This study will evaluate the effect of dexlansoprazole on bone homeostasis by assessing changes in biochemical markers of bone formation and bone resorption. This study will also assess changes in bone mineral density by dual-energy x-ray absorptiometry scan and other markers of bone homeostasis.

The study will consist of a 12-week screening period, a 26-week treatment period with a total of 5 visits during the treatment period and a follow-up visit at Week 52 for bone mineral density assessment.

ELIGIBILITY:
Inclusion Criteria:

* Is postmenopausal female in general good health with a body mass index of ≥18 and ≤30 kg/m2.
* Must have biochemical markers of bone formation, procollagen type 1 N-terminal propeptide and bone-specific alkaline phosphatase, and bone resorption, crosslinked β-C-terminal telopeptide of type 1 collagen and urine N-telopeptide within normal postmenopausal female ranges.
* Has not taken proton pump inhibitor medications within 6 months prior to screening and agrees to refrain from taking them through the last dose of study drug, except study-supplied dexlansoprazole or esomeprazole.

Exclusion Criteria:

* Has parathyroid hormone or thyroid stimulating hormone levels outside of the reference range at Week -12 and has 25-OH-D level <32 ng/mL at Week -2.
* Has baseline bone mineral density by dual-energy x-ray absorptiometry defined as a T-score lower than -2.0 at the total hip, spine, or femoral neck based on Caucasian reference values.
* Has a disorder strongly associated with osteoporosis
* Has a history of lumbar laminectomy, vertebroplasty, vertebral deformity or severe lumbar scoliosis that interferes with measurement or performance of the dual x-ray absorptiometry .
* Has a history or clinical manifestations of uncontrolled or significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, or psychiatric disorder as determined by the investigator which may affect the ability of the subject to participate or potentially confound the trial results.
* Has family history of genetic bone disorders.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2015-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (12):
- United States (12):
  - San Diego, California
  - Walnut Creek, California
  - Lakewood, Colorado
  - Hialeah, Florida
  - Jupiter, Florida
  - Bethesda, Maryland
  - Albuquerque, New Mexico
  - Spartanburg, South Carolina
  - Austin, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Hansen KE, Nieves JW, Nudurupati S, Metz DC, Perez MC. Dexlansoprazole and Esomeprazole Do Not Affect Bone Homeostasis in Healthy Postmenopausal Women. Gastroenterology. 2019 Mar;156(4):926-934.e6. doi: 10.1053/j.gastro.2018.11.023. Epub 2018 Nov 13. PMID 30445008
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 01 November 2010 (first subject signed informed consent form) to 1 February 2015.
Pre-assignment Details: Healthy post-menopausal women were enrolled equally in 1 of 3 treatment groups, once a day, placebo, 60 mg dexlansoprazole delayed-release capsules or 40 mg esomeprazole delayed-release capsules.
Groups:
- Esomeprazole 40 mg: Esomeprazole 40 mg, capsules, orally, once daily for up to 26 weeks. Participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 Ca 3 mg, intravenously and 44 Ca 8 mg, orally, once on Day-1 and Week 26.
Period: Main Study
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Started | 42 | 38 | 35
Safety Set: Received Study Drug | 41 | 38 | 35
Randomized, Not Treated | 1 | 0 | 0
Completed | 34 | 30 | 29
Not Completed | 8 | 8 | 6
Not completed — Adverse Event | 1 | 4 | 2
Not completed — Major Protocol Deviation | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Voluntary Withdrawal | 2 | 2 | 2
Not completed — Other Reason Not Specified | 0 | 1 | 1
Not completed — Randomized, Not Treated | 1 | 0 | 0
Period: Calcium Absorption Substudy
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Started | 14 | 10 | 10
Safety Set: Received Study Drug | 14 | 10 | 10
Completed | 12 | 8 | 10
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Major Protocol Deviation | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set includes all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg | Total
Number analyzed (Participants) | 41 | 38 | 35 | 114
Age, Continuous [Mean (Full Range); unit: years] — Population: Number analyzed are the participants with data available for Age
  years
    number analyzed (Participants) | 40 | 37 | 35 | 112
    (all) | 61.2 [51 to 73] | 62.4 [52 to 75] | 63.2 [54 to 74] | 62.2 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 35 | 114
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 11
  Not Hispanic or Latino | 38 | 33 | 32 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 37 | 34 | 33 | 104
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 38 | 35 | 114
Height [Mean (Full Range); unit: cm] | 164.4 [153 to 175] | 164.9 [154 to 178] | 164.6 [152 to 180] | 164.6 [152 to 180]
Weight [Mean (Full Range); unit: kg] | 69.25 [54.4 to 87.7] | 66.54 [51.4 to 92.0] | 69.47 [55.4 to 97.5] | 68.1 [51.4 to 97.5]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 25.61 [21.3 to 30.9] | 24.46 [18.2 to 31.3] | 25.65 [19.6 to 30.7] | 25.24 [18.2 to 31.3]
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 30 | 23 | 27 | 80
  Current smoker | 0 | 0 | 0 | 0
  Ex-smoker | 11 | 15 | 8 | 34
Alcohol Classification [Count of Participants; unit: Participants]
  Never drank | 6 | 6 | 6 | 18
  Current drinker | 30 | 31 | 27 | 88
  Ex-drinker | 5 | 1 | 2 | 8
Caffeine Consumption [Count of Participants; unit: Participants]
  Had caffeine consumption | 37 | 34 | 29 | 100
  Not had caffeine consumption | 4 | 4 | 6 | 14
Calcium at Screening Visit [Mean (Full Range); unit: mg/dL] | 9.93 [9.0 to 10.7] | 9.87 [9.0 to 10.7] | 9.97 [9.4 to 10.9] | 9.92 [9.0 to 10.9]
Vitamin D at Screening Visit [Mean (Full Range); unit: ng/mL] | 35.5 [13 to 74] | 33.2 [17 to 63] | 33.4 [11 to 75] | 34.1 [11 to 75]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 26 in Bone Formation Marker Aminoterminal Propeptide of Type 1 Collagen (P1NP)
Description: The percent change in bone formation marker P1NP measured at week 26 from P1NP measured at baseline. Serum samples for P1NP were analyzed at a central laboratory for bone biomarker P1NP using an electrochemiluminescence immunoassay measured in nanograms per milliliter (ng/mL).
Time Frame: Baseline and Week 26
Population: Participants from the Pharmacodynamic Set, all randomized participants who received study drug with evaluable calcium absorption data at Day 1 and Week 26, with data available for this outcome measure.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 32 | 31 | 26
percent change | -0.4 [-35 to 75] | 19.3 [-33 to 82] | 16.9 [-8 to 73]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 60 mg; Test type: Superiority or Other; Difference = 19.2, 95% CI 2-sided [7.0 to 30.2] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method
Statistical Analysis 2: Comparison: Placebo vs Esomeprazole 40 mg; Test type: Superiority or Other; Difference = 18.2, 95% CI 2-sided [6.7 to 30.4] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method

2. Primary Outcome: Percent Change From Baseline to Week 26 in Bone Resorption Marker C-telopeptide of Collagen Cross-links (CTX)
Description: The percent change in bone resorption marker CTX measured at week 26 from CTX measured at baseline. Plasma samples were analyzed at a central laboratory for bone biomarker CTX using an electrochemiluminescence immunoassay measured in ng/mL.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 32 | 31 | 26
percent change | 2.441 [-65.59 to 54.55] | 29.524 [-28.81 to 171.74] | 23.897 [-21.90 to 110.53]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 60 mg; Test type: Superiority or Other; Difference = 27.366, 95% CI 2-sided [12.749 to 42.957] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method
Statistical Analysis 2: Comparison: Placebo vs Esomeprazole 40 mg; Test type: Superiority or Other; Difference = 22.025, 95% CI 2-sided [8.357 to 35.714] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method

3. Secondary Outcome: Percent Change From Baseline to Week 26 in Urine N-telopeptide of Collagen Cross-links (NTx) Calculated
Description: The percent change in bone resorption marker NTx measured at week 26 from NTx measured at baseline. Urine samples were analyzed at a central laboratory for NTx using an enzyme-linked immunosorbent assay calculated as (nmol BCE/mmol creatinine). BCE=bone collagen equivalent
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 32 | 31 | 26
percent change | -6.1 [-53 to 86] | 16.9 [-45 to 100] | 6.2 [-45 to 67]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 60 mg; Test type: Superiority or Other; Difference = 20.1, 95% CI 2-sided [4.0 to 34.4] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method
Statistical Analysis 2: Comparison: Placebo vs Esomeprazole 40 mg; Test type: Superiority or Other; Difference = 11.6, 95% CI 2-sided [-2.7 to 28.3] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method

4. Secondary Outcome: Percent Change From Baseline to Week 26 in Bone-specific Alkaline Phosphatase (BsAP)
Description: The percent change in bone formation marker BsAP measured at week 26 from BsAP measured at baseline. Serum samples were analyzed at a central laboratory for bone biomarker BsAP using an enzyme immunoassay measured in units per liter (U/L).
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 32 | 31 | 26
percent change | 0.50 [-22.7 to 27.2] | 8.68 [-14.6 to 36.2] | 6.23 [-13.5 to 48.0]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 60 mg; Test type: Superiority or Other; Difference = 6.83, 95% CI 2-sided [0.40 to 12.78] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method
Statistical Analysis 2: Comparison: Placebo vs Esomeprazole 40 mg; Test type: Superiority or Other; Difference = 7.23, 95% CI 2-sided [0.59 to 12.86] — Difference estimated using Hodges-Lehmann estimation, and corresponding 95% CIs calculated using Moses method

5. Other Pre Specified Outcome: Percent Change From Baseline in P1NP at Week 13
Description: Serum samples for P1NP were analyzed using an electrochemiluminescence immunoassay measured in ng/mL.
Time Frame: Baseline and Week 13
Population: The pharmacodynamic set included participants from the safety set who had baseline and postbaseline values for any of the primary or secondary endpoints. The pharmacodynamic set where data for baseline and post-baseline assessments was available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 35 | 31 | 31
percent change | 6.7 (18.27) | 19.1 (25.02) | 11.6 (18.23)

6. Other Pre Specified Outcome: Percent Change From Baseline in CTX at Week 13
Description: Plasma samples were analyzed for bone biomarker CTX using an electrochemiluminescence immunoassay measured in ng/mL.
Time Frame: Baseline and Week 13
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 31 | 30
percent change | 7.510 (29.9739) | 32.069 (45.6413) | 23.212 (23.8900)

7. Other Pre Specified Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (BMD) Measured by Dual Energy X-ray Absorptiometry (DXA) at Week 26
Description: DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 26 | 27 | 24
percent change | -0.6632 (2.48314) | -1.6039 (2.58207) | -1.0596 (2.41731)

8. Other Pre Specified Outcome: Percent Change From Baseline in Total Hip BMD Measured by DXA at Week 26
Description: DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 26 | 27 | 24
percent change | -0.1928 (1.42242) | -0.7190 (1.78479) | -0.5330 (1.50491)

9. Other Pre Specified Outcome: Percent Change From Baseline in Lumbar Spine BMD Measured by DXA at Week 26
Description: DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 19 | 19 | 20
percent change | -0.2486 (3.29581) | -1.0753 (3.46909) | -1.2873 (2.06722)

10. Other Pre Specified Outcome: Percent Change From Week 26 in Femoral Neck BMD Measured by DXA at Week 52
Description: DXA is a means of measuring BMD through x-ray.
Time Frame: Week 26 and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 23 | 25 | 23
percent change | -0.0063 (2.57407) | -0.3439 (2.39680) | 0.2689 (2.67283)

11. Other Pre Specified Outcome: Percent Change From Weeks 26 in Total Hip BMD Measured by DXA at Week 52
Description: DXA is a means of measuring BMD through x-ray.
Time Frame: Week 26 and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 23 | 25 | 23
percent change | -0.0201 (1.28096) | -0.3324 (1.58091) | -0.0799 (1.81755)

12. Other Pre Specified Outcome: Percent Change From Weeks 26 in Lumbar Spine BMD Measured by DXA at Week 52
Time Frame: Week 26 and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 17 | 18 | 18
percent change | -0.4913 (3.01161) | -0.3561 (2.42934) | 0.8565 (2.46230)

13. Other Pre Specified Outcome: Number of Participants With Fracture Including Vertebral Fracture During Study Treatment
Time Frame: Baseline up to Week 26
Population: The pharmacodynamic set included participants from the safety set who had baseline and postbaseline values for any of the primary or secondary endpoints.
Measure: Number; unit: participants
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 38 | 36 | 34
participants | 0 | 0 | 0

14. Other Pre Specified Outcome: Change From Baseline in 24-hour Urinary Calcium Excretion at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram per day (mg/d)
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 29 | 29 | 24
milligram per day (mg/d)
  Baseline | 160.3 (76.16) | 184.8 (79.52) | 153.7 (90.09)
  Change at Week 26 | -24.4 (87.16) | -50.6 (84.95) | -49.7 (94.38)

15. Other Pre Specified Outcome: Change From Baseline in Parathyroid Hormone (PTH) at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 30 | 31
picogram per milliliter (pg/mL)
  Baseline | 30.67 (10.068) | 30.68 (11.917) | 31.10 (8.254)
  Change at Week 26: number analyzed (Participants) | 32 | 29 | 26
  Change at Week 26 | 2.16 (7.793) | 2.08 (7.765) | 3.37 (9.525)

16. Other Pre Specified Outcome: Change From Baseline in Serum Calcium at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 32 | 30
milligram per deciliter (mg/dL)
  Baseline | 9.48 (0.347) | 9.47 (0.291) | 9.58 (0.308)
  Change at Week 26: number analyzed (Participants) | 32 | 31 | 26
  Change at Week 26 | -0.03 (0.440) | -0.03 (0.333) | -0.07 (0.331)

17. Other Pre Specified Outcome: Change From Baseline in Serum Phosphorus at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 32 | 30
mg/dL
  Baseline | 3.73 (0.377) | 3.92 (0.422) | 3.89 (0.335)
  Change at Week 26: number analyzed (Participants) | 32 | 31 | 26
  Change at Week 26 | 0.08 (0.445) | 0.07 (0.271) | 0.03 (0.393)

18. Other Pre Specified Outcome: Change From Baseline in Serum Magnesium at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliequivalent per liter (meq/L)
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 32 | 30
milliequivalent per liter (meq/L)
  Baseline | 1.72 (0.124) | 1.72 (0.145) | 1.77 (0.127)
  Change at Week 26: number analyzed (Participants) | 32 | 31 | 26
  Change at Week 26 | -0.01 (0.118) | -0.02 (0.109) | -0.03 (0.096)

19. Other Pre Specified Outcome: Change From Baseline in Urine Magnesium at Week 26
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: meq/L
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 35 | 32 | 31
meq/L
  Baseline | 3.8 (2.11) | 4.6 (3.46) | 4.1 (2.85)
  Change at Week 26: number analyzed (Participants) | 31 | 31 | 26
  Change at Week 26 | -0.1 (2.41) | -0.8 (2.83) | -0.5 (2.80)

20. Other Pre Specified Outcome: Change From Baseline to Week 26 in Vitamin D3 (25-OH-D) Level
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 36 | 32 | 31
ng/mL
  Baseline | 41.3 (9.96) | 39.4 (11.64) | 36.4 (8.48)
  Change at Week 26: number analyzed (Participants) | 32 | 30 | 26
  Change at Week 26 | -2.7 (10.20) | -0.6 (12.07) | 1.1 (9.75)

21. Other Pre Specified Outcome: Change From Baseline in Intestinal Calcium Absorption by True Fractional Calcium Absorption (TFCA) in a Subset of Participants at Week 26
Time Frame: Baseline and Week 26
Population: The PD set included participants from the safety set who had baseline and postbaseline values for any of the primary or secondary endpoints. The PD set included participants with evaluable calcium absorption data on Day-1 and Week 26.
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40 mg
Number analyzed (Participants) | 12 | 9 | 10
mg/d
  Baseline | 0.18 (0.064) | 0.18 (0.043) | 0.17 (0.049)
  Change at week 26 | -0.01 (0.049) | 0.02 (0.042) | 0.05 (0.050)

ADVERSE EVENTS:
Time Frame: First dose of study drug and within 30 days of the last dose of study drug (Up to 30 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Placebo: Placebo-matching capsules, orally, once daily for up to 26 weeks.
- Dexlansoprazole 60 mg: Dexlansoprazole 60 mg, capsules, orally, once daily for up to 26 weeks.
- Esomeprazole 40mg: Esomeprazole 40 mg, capsules, orally, once daily for up to 26 weeks.
- Calcium Absorption Sub Study: Placebo: Following the main study participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 calcium (42 Ca) 3 milligram (mg), intravenously and 44 calcium (44 Ca) 8 mg, orally, once on Day-1 and Week 26.
- Calcium Absorption Sub Study: Dexlansoprazole 60 mg; Calcium Absorption Sub Study: Esomeprazole 40 mg: Following the main study Participants had the option to participate in the calcium absorption sub study to receive calcium isotope 42 Ca 3 mg, intravenously and 44 Ca 8 mg, orally, once on Day-1 and Week 26.
Arm/Group | Placebo | Dexlansoprazole 60 mg | Esomeprazole 40mg | Calcium Absorption Sub Study: Placebo | Calcium Absorption Sub Study: Dexlansoprazole 60 mg | Calcium Absorption Sub Study: Esomeprazole 40 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38 | 0/35 | 0/14 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/38 | 0/35 | 0/14 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/41 | 8/38 | 9/35 | 3/14 | 4/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Dexlansoprazole 60 mg (N=38) | Esomeprazole 40mg (N=35) | Calcium Absorption Sub Study: Placebo (N=14) | Calcium Absorption Sub Study: Dexlansoprazole 60 mg (N=10) | Calcium Absorption Sub Study: Esomeprazole 40 mg (N=10)
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Dexlansoprazole 60 mg (N=38) | Esomeprazole 40mg (N=35) | Calcium Absorption Sub Study: Placebo (N=14) | Calcium Absorption Sub Study: Dexlansoprazole 60 mg (N=10) | Calcium Absorption Sub Study: Esomeprazole 40 mg (N=10)
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1 | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.